CLINICAL TRIAL: NCT03300908
Title: Contextualizing & Responding to HIV Risk Behaviors Among Black Drug Offenders
Brief Title: Contextualizing & Responding to HIV Risk Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tawandra Rowell-Cunsolo, Assistant Professor of Social Welfare Science, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAL7007; K01DA036411 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — omega-Chloroacetophenone

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to Project ADHERE, or the control condition, MACE. The randomization process was described to participants during the informed consent process.
Who Masked: Participant
Masking Description: Participants were not aware of which intervention they were assigned to. A randomization scheme was developed and participants were assigned to treatment groups accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project ADHERE (Experimental): Participants will receive a 3-session antiretroviral medication adherence and risk reduction intervention called Project ADHERE.
  Interventions: Behavioral: Project ADHERE
- Control MACE (Active Comparator): Participants will receive a one-session antiretroviral medication adherence intervention called MACE.
  Interventions: Behavioral: MACE

INTERVENTIONS:
Behavioral: Project ADHERE — This is a 3-session ART medication adherence and risk reduction intervention. Participants are educated about the importance of staying healthy and taking their medication as prescribed; to discuss importance of improved immune functioning and what their "viral load" means; reminded that they can still infect others with HIV, and that there currently is no cure for HIV; expected to generate strategies to overcome adherence barriers; educated about sexually transmitted infections (STI)/HIV transmission modes; assisted in devising an appropriate medication adherence and risk reduction plan. Participants will report their progress and discuss challenges experienced when implementing their medication adherence and risk reduction plans while establishing short- and long-term goals.
  Other Names: Project ADHerence Education and Risk Evaluation
  Arms: Project ADHERE
Behavioral: MACE — This one-session medication adherence intervention covers the following content: 1) a discussion on what viral load represents and what HIV does to the body; 2) referral to a provider for participants without a provider; 3) the importance of maintaining regular contact with a health care provider; and 4) benefits of being retained in care.
  Other Names: Medication Adherence and Care Engagement
  Arms: Control MACE

SUMMARY:
The purpose of this study was to pilot test the potential for improvement in antiretroviral medication adherence of a an adapted group-based, multi-session, community-based Antiretroviral Therapy (ART) adherence and risk reduction intervention, Project ADHerence Education and Risk Evaluation (ADHERE). Project ADHERE was compared to a single-session group-based medication adherence intervention, Medication Adherence and Care Engagement (MACE).

A secondary aim was to examine the impact of Project ADHERE on HIV risk behaviors (i.e., illicit drug use and unprotected sexual behavior).

This study was designed to inform, design, and pilot test the two antiretroviral medication adherence interventions for HIV-infected formerly incarcerated individuals.

DETAILED DESCRIPTION:
Formerly incarcerated Black drug offenders are at an elevated risk for HIV infection. Despite substantial research expressing the need for HIV prevention services for ex-offenders postrelease, this population has limited access to quality programming and services related to HIV risk reduction. This K01 application seeks to inform and adapt an HIV risk reduction intervention to address the needs of formerly incarcerated Black drug offenders who are being released from prisons in the New York City metropolitan area.The study will utilize qualitative and quantitative methods to inform and adapt an HIV prevention intervention for this study population.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. HIV seropositive with "detectable" viral load (VL)(defined as >50 copies/mL)
3. history of drug use (used illicit drugs within the past year)
4. experienced incarceration in prison or jail within the past five years

Exclusion Criteria:

1. living in a healthcare or assisted living facility
2. experienced incarceration longer than five years ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants who reached at least 85% medication adherence rate. | Over a 3-month period
  Self-report data and viral loads to test for medication adherence will be collected and analyzed to yield the rate (%).

SECONDARY OUTCOMES:
Percentage of participants with HIV risk behaviors | Over a 3-month period
  Information on illicit drug use and unprotected sexual behavior wil be collected and analyzed. We sought to reduce the frequency of illicit drug use, and instance of unprotected sexual behavior as calculated in the percentage of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tawandra Rowell-Cunsolo, MD, Principal Investigator — Assistant Professor of Social Welfare Science (in Nursing), Nursing Scholarship & Research
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided